CLINICAL TRIAL: NCT03832257
Title: AHRQ Health Services Research Projects: Making Health Care Safer in Ambulatory Care Settings and Long Term Care Facilities
Brief Title: Improving Safety of Transitions to Skilled Nursing Care Using Videoconferencing
Acronym: ECHO-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brown University (Other); Hebrew SeniorLife (Other)
Responsible Party: Principal Investigator, Lewis Lipsitz, Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P000457
Record Dates: First submitted 2019-02-03; First posted 2019-02-06 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Acute Disease
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECHO CT Intervention (Experimental): Weekly video conference between hospitalist at Beth Israel and skilled nursing facilities.
  Interventions: Other: ECHO CT Intervention
- Matched Non- Participating Facilities (Other): Matched non-participating facilities
  Interventions: Other: Matched Non-Participating Facilities

INTERVENTIONS:
Other: ECHO CT Intervention — weekly video conference between hospitalist and skilled nursing facilities
  Arms: ECHO CT Intervention
Other: Matched Non-Participating Facilities — Matched Non-Participating Facilities
  Arms: Matched Non- Participating Facilities

SUMMARY:
This prospective cohort study seeks to determine if the ECHO-CT program, a healthcare videoconferencing program, can improve clinical outcomes while reducing cost and resource utilization when expanded to a community hospital setting. Data will be analyzed on the facility level and patient level.

DETAILED DESCRIPTION:
ECHO-Care Transitions is a healthcare outreach program utilizing videoconferencing technology to improve the quality and efficiency of care transitions for medically-complex elderly patients by connecting post-acute care facilities that receive BIDMC patients with a multidisciplinary BIDMC team that sends these patients following discharge. This case-control study seeks to determine if ECHO-CT can improve clinical outcomes and reduce cost and resource utilization during transitions of care in both an academic (BIDMC Boston) and community (BIDMC Needham) hospital.

Our prospective cohort study of the ECHO-CT intervention will take place in the two Boston-area hospitals, one providing tertiary care and one community-based care, in which the outcomes of patients transferred to Skilled Nursing Facilities (SNFs) associated with these hospitals will be compared to those transferred to SNFs from similar hospitals in New England. We will also be comparing outcomes from individual patients enrolled in the ECHO program to matched controls. Using a national database available from the Brown University Center for Gerontology and Healthcare Research, the outcomes of Medicare beneficiaries residing in SNFs that are participating in ECHO-CT will be compared to those in the comparison group using a difference-of-difference analytic approach. Analyses will be adjusted for potential confounders as appropriate.

In this study, the investigators also plan to measure satisfaction as well as process, utilization, cost and patient safety outcomes to determine best practices for implementing the program at a community hospital and affiliated SNFs.

Data will be obtained from the following sources:

1. Protected health information (PHI) from resident assessment data, as well as Medicare claims and enrollment data to be obtained via a data use agreement (DUA) with the Centers for Medicare and Medicaid Services (CMS) by the Brown University Center for Gerontology and Health Care Research during years 2-3 of the study to include the following:

   1. The resident Minimum Data Set Resident Assessment (MDS) assessments. The MDS has nearly 400 data elements including cognitive function, communication/hearing problems, physical functioning, continence, psycho-social well-being, mood state, activity and recreation, diagnoses, health conditions, nutritional status, oral/dental status, skin conditions, special treatments, and medication use. The assessments are done for all patients admitted to Medicare and Medicaid certified SNFs, including enrollees in both traditional Medicare and Medicare Advantage. These data will already be housed at Brown University,Brown has an active DUA to obtain quarterly pulls of the population of MDS assessments .
   2. Medicare claims which will be used to ascertain 30-day costs, re-hospitalizations, and use of other medical services by Medicare fee for service (FFS) patients admitted to the SNFs. The data also include diagnosis fields to ascertain comorbidities.
   3. Medicare enrollment file includes demographic information such as sex and race, dates of birth and death, and various indicators of Medicare/Medicaid eligibility, Part D eligibility, and Medicare Advantage enrollment.
   4. BIDMC will collect and share ECHO-CT participating patient's social security number and health insurance claims number with Brown University. Their clinical information will be matched with control patients from the Medicare claims data to show study effect on 30-day costs, re-hospitalizations rate and patient length of stay.
2. In addition to aggregates derived from above, facility level data will come from the Certification and Survey Provider Enhanced Reporting (CASPER) data, which are publicly available and based upon facility surveys for Medicare/Medicaid certification. They will be used in addition to data from "Nursing Home Compare and the Long Term Care: Facts on Care in the US (LTCFocus.org) websites to describe the SNFs.
3. Intervention-specific data: Project-specific quality improvement data derived from questionnaires, staff satisfaction surveys, and structured meeting minutes will be designed and evaluated by BIDMC and Hebrew Senior Life

   1. SNF Satisfaction: Every 6 months the investigators will send a satisfaction questionnaire to the hospitals and SNFs participating in ECHO-CT to assess their views of the ECHO-CT sessions, the value of time spent, feelings of empowerment, inter-professional relationships, learning, and recommendations. All answers to the survey questions will be kept strictly confidential. This information will be used to improve the content and organization of the sessions and to develop tools for dissemination (Aim 3). The investigators will develop the satisfaction questionnaire during the first 6 months of the project, building upon our previous survey experience and literature review. Metrics to quantify the quality of transitional care will be derived from the work of Coleman et al.3 and incorporated into the questionnaire. Survey design and evaluation will be conducted by the outcome evaluation group under the leadership of Dr. Thomas Travison at Hebrew SeniorLife's Institute for Aging Research.
   2. Process assessment: The investigators will keep attendance logs to assess adherence to the ECHO-CT intervention and its changes over time. Any consistent decline in staff attendance for 2 or more weeks will be followed up by phone calls to assess barriers to participation and corrective actions will be taken. These may include changing to a more convenient time, identifying other providers who can attend instead, contacting facility administrators or medical directors for their support, and providing incentive gifts or continuing education credits In addition, during each ECHO-CT session, the hospital based team will inquire about unexpected outcomes or issues that arose during the transition process, including those related to patients already discussed. This element will allow for an ongoing technology-enabled learning platform and continuous quality improvement mechanism over the course of the proposed project. The value of the video-conferencing approach is that it creates a mutually trusting learning community in which "all teach and all learn."

ELIGIBILITY:
Facility Inclusion Criteria:

* SNF receives approximately the middle third of referral volume (approx. 20-100 referrals/ average 40 per year)
* SNF not so highly engaged with acute hospital that their patients are less likely to benefit from the intervention.
* SNF affiliated with BIDMC Boston or BIDMC Needham

Facility Exclusion Criteria:

* Has not recently participated in ECHO CT
* Do not send anyone to ECHO CT training
* Clinicians are unwilling to make a commitment to attend at least 75% of video conferences

Patient Selection:

ECHO-CT Group:

Inclusion Criteria: Patients that were discharged from BIDMC and admitted to skilled nursing facilities that are participating in ECHO-CT between April 2019 and March 2021.

Exclusion Criteria: Patients discharged from a hospital other than BIDMC. Patients admitted to a skilled nursing facility that is not participating in ECHO-CT.

Control Group:

Inclusion Criteria: Patients from skilled nursing facilities not participating in ECHO.

Exclusion Criteria: Patients discharged from BIDMC to one of our participating SNFs during the study period of April 2019- March 2021

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10708 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
30-Day Readmission Rates | 30-Days
  Number of hospital readmissions over 30 day period among participating SNF sites

SECONDARY OUTCOMES:
Health Care Utilization | up to 90 days
  Includes average length of stay in the facility
Health Care Cost | 30-days
  Total 30-day Medicare costs for fee-for-service patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora S, Thornton K, Jenkusky SM, Parish B, Scaletti JV. Project ECHO: linking university specialists with rural and prison-based clinicians to improve care for people with chronic hepatitis C in New Mexico. Public Health Rep. 2007;122 Suppl 2(Suppl 2):74-7. doi: 10.1177/00333549071220S214. PMID 17542458
- [Background] Arora S, Thornton K, Murata G, Deming P, Kalishman S, Dion D, Parish B, Burke T, Pak W, Dunkelberg J, Kistin M, Brown J, Jenkusky S, Komaromy M, Qualls C. Outcomes of treatment for hepatitis C virus infection by primary care providers. N Engl J Med. 2011 Jun 9;364(23):2199-207. doi: 10.1056/NEJMoa1009370. Epub 2011 Jun 1. PMID 21631316
- [Background] Boltz M, Parke B, Shuluk J, Capezuti E, Galvin JE. Care of the older adult in the emergency department: nurses views of the pressing issues. Gerontologist. 2013 Jun;53(3):441-53. doi: 10.1093/geront/gnt004. Epub 2013 Feb 26. PMID 23442380
- [Background] Coleman EA, Berenson RA. Lost in transition: challenges and opportunities for improving the quality of transitional care. Ann Intern Med. 2004 Oct 5;141(7):533-6. doi: 10.7326/0003-4819-141-7-200410050-00009. PMID 15466770
- [Background] Kessler C, Williams MC, Moustoukas JN, Pappas C. Transitions of care for the geriatric patient in the emergency department. Clin Geriatr Med. 2013 Feb;29(1):49-69. doi: 10.1016/j.cger.2012.10.005. PMID 23177600
- [Background] Moore AB, Krupp JE, Dufour AB, Sircar M, Travison TG, Abrams A, Farris G, Mattison MLP, Lipsitz LA. Improving Transitions to Postacute Care for Elderly Patients Using a Novel Video-Conferencing Program: ECHO-Care Transitions. Am J Med. 2017 Oct;130(10):1199-1204. doi: 10.1016/j.amjmed.2017.04.041. Epub 2017 May 25. PMID 28551043
- [Background] Marks C, Loehrer S, McCarthy D. Hospital readmissions: measuring for improvement, accountability, and patients. Issue Brief (Commonw Fund). 2013 Sep;24:1-8. PMID 24044140
- [Background] Mor V, Intrator O, Feng Z, Grabowski DC. The revolving door of rehospitalization from skilled nursing facilities. Health Aff (Millwood). 2010 Jan-Feb;29(1):57-64. doi: 10.1377/hlthaff.2009.0629. PMID 20048361
- [Background] LaMantia MA, Scheunemann LP, Viera AJ, Busby-Whitehead J, Hanson LC. Interventions to improve transitional care between nursing homes and hospitals: a systematic review. J Am Geriatr Soc. 2010 Apr;58(4):777-82. doi: 10.1111/j.1532-5415.2010.02776.x. PMID 20398162
- [Background] Austin BJ. Rehospitalization from skilled nursing facilities: implications for policy. Find Brief. 2010 Feb;12(9):1-3. PMID 20222212
- [Background] Ouslander JG, Diaz S, Hain D, Tappen R. Frequency and diagnoses associated with 7- and 30-day readmission of skilled nursing facility patients to a nonteaching community hospital. J Am Med Dir Assoc. 2011 Mar;12(3):195-203. doi: 10.1016/j.jamda.2010.02.015. Epub 2010 Aug 12. PMID 21333921